CLINICAL TRIAL: NCT02088255
Title: Walking Training With Partial Body Weight Support on Static and Dynamic Surfaces in Individuals With Hemiparesis Due to Stroke
Brief Title: Walking Training With Partial Body Weight Support on Static and Dynamic Surfaces in Stroke Survivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cruzeiro do Sul (Other)
Responsible Party: Principal Investigator, Gabriela Lopes Gama, Principal Investigator, Universidade Cruzeiro do Sul
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CE/UCS-016/2013
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2015-07

CONDITIONS: Stroke
Keywords: Rehabilitation; Gait; Stroke; Biomechanics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Static surface (Active Comparator): The subjects will do the walking training with partial body weight support on static surface. The will be submitted to three weekly training sessions of approximately 45 minutes each , for six weeks , totaling 18 sessions
  Interventions: Procedure: Static surface
- dynamic surface (Active Comparator): The subjects will do the walking training with partial body weight support on dynamic surface. The will be submitted to three weekly training sessions of approximately 45 minutes each , for six weeks , totaling 18 sessions
  Interventions: Procedure: Dynamic surface

INTERVENTIONS:
Procedure: Static surface — During all session time the subject will walk on the floor with partial body weight support. This protocol will be repeated in all sessions.
  Other Names: floor walking training
  Arms: Static surface
Procedure: Dynamic surface — During all session time the subject will walk on the treadmill with partial body weight support. This protocol will be repeated in all sessions.
  Other Names: Treadmill Training
  Arms: dynamic surface

SUMMARY:
The purpose of this study is evaluate the effects of walking training with partial body weight support on static (floor) and dynamic (treadmill) surfaces in individuals with hemiparesis due to stroke. For this purpose, two training protocols will be employed in three experimental groups: G1 will do the walking training with partial body weight support on static surfaces and G2 will do the walking training with partial body weight support on dynamic surfaces

ELIGIBILITY:
Inclusion Criteria:

* One-sided hemiparesis, No heart disease (or medical clearance to participate in the study), No orthopedic impairments and / or neurological symptoms that may alter the the gait, no history of thrombophlebitis or deep vein thrombosis, Ability to understand and follow verbal commands, Can walk alone or with canes of approximately 10 m; Spasticity degree mild to moderate in the affected lower limb with levels of classification between 0 and 2 in the Ashworth spasticity scale modified

Exclusion Criteria:

* Heart frequency increase more than 75% of the maximum or have any other general instability during training that may lead risk for the health during the training,

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the gait velocity | Baseline, immediately after and six weeks after training cessation.
  Speed at which subjects walked measured by the 10 meters test

SECONDARY OUTCOMES:
Distribution of body weight | Baseline, immediately after and six weeks after training cessation.
  Body weight Distribution measured while subjects are in a static position on two force platforms.
Functional independence | Baseline, immediately after and six weeks after training cessation.
  a score was assigned for each everyday activity, according to the amount of assistance required to perform it. Measured by a clinical scale (Functional Independence Measure Scale.
Lower limb recovery | Baseline, immediately after and six weeks after training cessation.
  Measured by a clinical scale (Fulgy Meyer).
Endurance | Baseline, immediately after and six weeks after training cessation.
  Measured by the 6 minutes walking test

OTHER OUTCOMES:
Spacial and temporal variables | Baseline, immediately after and six weeks after training cessation.
  Measured while subjects are walking at a comfortable speed
Center of Pressure | Baseline, immediately after and six weeks after training cessation.
  Behavior of the Center of Pressure in gait and gait initiation measured by the force plates during the gait and gait initiation. Center of Pressure distance and seed displacement will be measured during the task.
articular and segment angles | Baseline, immediately after and six weeks after training cessation.
  Measured while subjects are walking at a comfortable speed

CONTACTS AND LOCATIONS:
Locations (1):
- Cruzeiro do Sul University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gama GL, Celestino ML, Barela JA, Forrester L, Whitall J, Barela AM. Effects of Gait Training With Body Weight Support on a Treadmill Versus Overground in Individuals With Stroke. Arch Phys Med Rehabil. 2017 Apr;98(4):738-745. doi: 10.1016/j.apmr.2016.11.022. Epub 2016 Dec 27. PMID 28034719